CLINICAL TRIAL: NCT05225012
Title: Providing Emotional Support Around the Point of Multiple Sclerosis Diagnosis: PrEliMS 2
Acronym: PrEliMS2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21082
Record Dates: First submitted 2022-01-10; First posted 2022-02-04 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Multiple Sclerosis
Keywords: Acceptance and Commitment Therapy
MeSH Terms: conditions — Multiple Sclerosis | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Intervention Model Description: Case series design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PrEliMS Intervention (Experimental): We will ask participants to complete the psychological impact of MS scale, anxiety/depression questionnaires and visual analogue scales once a week throughout their involvement in the study (estimated to be 9 weeks). The baseline will be established over a period of the first three weeks (before participants start the intervention). Participants will also be asked to complete a second set of questionnaires (secondary measures) before starting the intervention, to assess quality of life, stress, the impact of MS, MS-related self-efficacy and fatigue.
  Participants will then be invited to an optional semi-structured, feedback interview to provide qualitative information on their experience of the intervention.
  Interventions: Other: Acceptance and Commitment Therapy

INTERVENTIONS:
Other: Acceptance and Commitment Therapy — Participants will then commence the intervention for the next 4 weeks. They will be sent the workbook via post. This will not be a standalone self-help intervention; participants will progress through the workbook alongside weekly emotional support sessions. These will either be over the phone or using an online video-call software, depending on participants preference. The first session will be an hour long to set-up the workbook, answer questions and go through goal setting. The following three weekly sessions will be half an hour to revisit exercises in the workbook, answer questions and review how the workbook progress is going. All sessions will be delivered by a trainee clinical psychologist who will receive standardised training and ongoing supervision from an experienced clinical psychologist.

SUMMARY:
Emotional support following Multiple Sclerosis (MS) diagnosis is not part of the current service provision. However, research has identified a need for this as poor adjustment to diagnosis has been linked to higher levels of psychological distress. A previous study, named 'Providing Emotional Support Around the Point of MS Diagnosis' (PrEliMS), explored how best to provide support. People with MS completed a self-help workbook, alongside receiving support from MS nurses. The workbook is based on a psychological therapy called Acceptance and Commitment Therapy and was developed through focus groups of people with MS, relevant stakeholders, and clinical expertise. In this study, issues were found with parts of the workbook content and delivery. Nurses found it difficult to facilitate this alongside their usual MS Nurse care and felt psychological distress was not within their remit.

In this study, the investigators will

* explore how effective the PrEliMS workbook is at reducing distress from MS diagnosis, when delivered by a Psychology Practitioner (Trainee Clinical Psychologist)
* compare delivery by a Psychology Practitioner with the data from the Nurse delivered PrEliMS trial to explore which is more effective
* explore experience of the PrEliMS-2 intervention and potential improvements.

The investigators will recruit between three and seven people from an MS clinic who have received an MS diagnosis in the last year and consent to taking part. Participants will meet with a Psychology Practitioner (over the phone or online) once a week for four weeks, alongside completing the workbook. The investigators will also ask participants to complete questionnaires to examine their levels of psychological distress. Interviews will then be conducted to get feedback for refining the workbook.

The overall study will last a year

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 and/or over.
2. Received a new diagnosis of MS within the last twelve months, confirmed by a Consultant Neurologist.
3. Scores ≥18 on the MSIS-Psy.

Exclusion Criteria:

1. Unable or willing to give informed consent.
2. Individuals currently receiving psychological therapy, to ensure any change cannot be attributed to another intervention.
3. Individuals who have had a prior diagnosis of psychological distress, e.g., Depression or Anxiety Disorder, to ensure participants are as homogenous as possible. The intervention is aimed at distress specifically related to receiving an MS diagnosis.
4. Unable to speak and read English (as all measure used have been standardised and validated in English, and the workbook is only available in English).
5. Unable to use/do not have access to a telephone or a computer with internet connection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2022-08-12 (Actual); Primary Completion 2023-04-28 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Perceived psychological impact of MS | Once a week from baseline to 1-week follow-up, and 1-month follow-up
  The principle primary outcome (main primary outcome of interest). Multiple Sclerosis Impact Scale-Psychological Subscale (MSIS-29-PSYCH; Hobart et al., 2001; Ramp et al., 2009). Total scores range from 0-45, with higher scores indicating greater perceived psychological impact of MS. Nine scaled questions with scale values ranging from 1-5.
Patient Health Questionnaire - 9 (PHQ-9) | Once a week from baseline to 1-week follow-up, and 1-month follow-up
  Change in the level of depression symptoms. Higher scores indicate a worse outcome, total scores range from 0-27, scale values range from 0-3.
Generalised Anxiety Disorder - 7 (GAD-7) | Once a week from baseline to 1-week follow-up, and 1-month follow-up
  Change in the level of anxiety symptoms. Higher scores indicate a worse outcome, total scores range from 0-21, scale values range from 0-3.
Visual Analogue Scales | Once a week from baseline to 1-week follow-up, and 1-month follow-up
  Change in (1) the level of psychological distress related to receiving an MS diagnosis, (2) confidence in managing the physical impact day to day and (3) confidence in managing the psychological impact day to day. Scale ranges from 0-10.

SECONDARY OUTCOMES:
Health-related quality of life | Baseline, 1-week follow-up and 1-month follow-up
  EQ-5D-5L (Herdman et al., 2011). Five scaled questions assessing five domains of quality of life (mobility, self-care, usual activities, pain/discomfort, anxiety/depression. Each response corresponds to a 1-digit number. The total responses are combined into a 5-digit number to represent health state, e.g., 11111 represents no problems in health state. These are then converted to an index score; higher scores indicate greater health related quality of life.
Perceived levels of stress | Baseline, 1-week follow-up and 1-month follow-up
  Perceived Stress Scale 4 (PSS4; Cohen et al., 1983). Total scores range from 0-40, with higher scores indicating greater perceived level of stress. Ten scale questions, scaled values range from 0-4.
Self efficacy in the context of MS | Baseline, 1-week follow-up and 1-month follow-up
  Multiple Sclerosis Self Efficacy Scale (MSSES; Rigby et al., 2003). Total score ranges from 0-84, with higher scores indicating greater level of self-efficacy. 14 scaled questions with values ranging from 1-6.
Levels of fatigue | Baseline, 1-week follow-up and 1-month follow-up
  Modified Impact Fatigue Scale; abbreviated version (MFIS-5; Fisk et al., 1994; Fischer et al., 1999). Total score ranges from 0-20; higher scores indicate greater impact of fatigue. Scale scores range from 0-4 with 5 scaled questions.

OTHER OUTCOMES:
Comprehensive Assessment of Acceptance and Commitment Therapy processes (CompACT-8; Morris, 2019; Dawson & Golijani-Moghaddam, 2020). | Once a week from baseline to 1-week follow-up, and 1-month follow-up
  Process measure. Scale to measure change in ACT-process of psychological flexibility. Higher scores indicate a better outcome, total scores range from 0-48, scale values range from 0-6.

CONTACTS AND LOCATIONS:
Overall Officials: Nima Moghaddam, DClinPsy, Study Chair — University of Lincoln; Nikos Evangelou, DPhil, Principal Investigator — University of Nottingham
Locations (1):
- Queens Medical Hospital, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No